CLINICAL TRIAL: NCT01873378
Title: Surgical Effects of GnRH Agonist Pretreatment on Cold Loop Hysteroscopic Myomectomy.
Brief Title: GnRH Agonist Pretreatment in Hysteroscopic Myomectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera S. Maria della Misericordia (Other)
Responsible Party: Principal Investigator, Sandro Gerli, Assistant Professor, Azienda Ospedaliera S. Maria della Misericordia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GnRHa hysteroscopic myomectomy
Record Dates: First submitted 2013-06-01; First posted 2013-06-10 (Estimated); Last update posted 2015-08-11 (Estimated); Status verified 2015-08

CONDITIONS: Uterine Myoma
Keywords: Uterine myoma; GnRHa; Hysteroscopy; Cold loop
MeSH Terms: conditions — Myofibroma | interventions — Triptorelin Pamoate

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- GnRH agonist pretreatment (Experimental): triptorelin 3.75 mg, im, monthly, three times
  Interventions: Drug: Triptorelin 3.75 mg
- No pharmacological treatment (No Intervention)

INTERVENTIONS:
Drug: Triptorelin 3.75 mg
  Arms: GnRH agonist pretreatment

SUMMARY:
The primary outcome of this study is to assess if the GnRHa administration before cold loop hysteroscopic myomectomy contributes to accomplish the treatment in only one surgical procedure. Moreover, we will investigate the intraoperative influence of such pharmacologic therapy in terms of distension liquid absorption and duration of the procedures.

ELIGIBILITY:
Inclusion Criteria:

* submucous myoma diagnosed by vaginal ultrasonography and confirmed by diagnostic hysteroscopy
* premenopausal status

Exclusion Criteria:

* present or past history of cancer
* pregnancy
* presence of associated multiple polyps
* presence of > 2 myomas
* associated nonhysteroscopic surgical procedures

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2013-01; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
To assess if the GnRHa administration before cold loop hysteroscopic myomectomy contributes to accomplish the treatment in only one surgical procedure. | Just finished the surgical procedure.

SECONDARY OUTCOMES:
Minutes (surgical procedure time), milliliters (fluid absorption during the procedure). | Just finished the surgical procedure.

CONTACTS AND LOCATIONS:
Overall Officials: sandro gerli, MD, Principal Investigator — University of Perugia, Perugia, Italy
Locations (1):
- Arbor Vitae Endoscopic Centre, Rome, Italy, Italy

REFERENCES:
- [Derived] Favilli A, Mazzon I, Grasso M, Horvath S, Bini V, Di Renzo GC, Gerli S. Intraoperative Effect of Preoperative Gonadotropin-Releasing Hormone Analogue Administration in Women Undergoing Cold Loop Hysteroscopic Myomectomy: A Randomized Controlled Trial. J Minim Invasive Gynecol. 2018 May-Jun;25(4):706-714. doi: 10.1016/j.jmig.2017.11.011. Epub 2017 Nov 24. PMID 29180306